CLINICAL TRIAL: NCT04929964
Title: COVID 19 Pandemic: Effect on Management of Patients With Breast Cancer; Single Center Study
Brief Title: COVID-19 Pandemic: Effect on Management of Patients With Breast Cancer
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Mehwish Mooghal , MBBS (Other)
Responsible Party: Sponsor-Investigator, Mehwish Mooghal , MBBS, Resident Surgery at PNS Shifa Hospital Karachi, Bahria University
Organization: Bahria University (Other)
Other Study IDs: COV-19 BUMDC
Record Dates: First submitted 2021-06-13; First posted 2021-06-18 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Breast Cancer Stage; Isolation, Social; Locally Advanced Breast Cancer
Keywords: Breast Cancer; Covid-19; Modified Radical Mastectomy; Breast Conservation Surgery
MeSH Terms: conditions — COVID-19; Social Isolation; Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer
  Interventions: Procedure: MRM , Toilet Mastectomy , BCS

INTERVENTIONS:
Procedure: MRM , Toilet Mastectomy , BCS — MRM , modified radical mastectomy : removing breast and axilla toilet mastectomy : palliative removal of tumor load BCS ,Breast conservative surgery

SUMMARY:
The objective was to find out the impact of COVID-19 on stage of breast cancer at presentation and its effects on overall onco-surgical management. The investigator carried out this research to see the presenting stage of breast cancer in the participants in this pandemic and correlate its effect on stage of breast cancer and upstaging of disease

DETAILED DESCRIPTION:
This retrospective observational study was conducted at department of surgery PNS Shifa hospital Karachi after obtaining permission from ethical review committee. Participant's data of all operated cases for suspicious lump breast (abnormal findings on ultrasound and mammogram, BIRAD III or above and abnormal FNAC results;C3 or above) from January1,2020 to 31 January 2021 was retrieved. Out of these only those participants were included in whom the diagnosis of breast cancer was confirmed on histo-pathological examination. Participants who had already had their surgery pre covid (December 2019), were excluded. Data were collected on standard pre-designed questionnaire and from paper documents retrieved from patient records. Participant presentation time was calculated as the time interval between the appearance of the first symptoms of breast cancer (day 0) and the date of initial presentation to hospital by patient and consultation for breast symptoms. Time taken for start of treatment was calculated by counting number of days from the first presentation day to hospital until the date when definitive treatment for Carcinoma Breast was initiated (chemo/radio/surgery). Time duration for definitive surgery was counted from the day of first presentation to the hospital till the date surgery was conducted(modified radical mastectomy (MRM)/breast conserving surgery (BCS)/toilet mastectomy).

Presentation 'Delay' was defined as a patient reporting to the hospital for medical advice 30 days after noticing the first possible symptoms of breast cancer while time taken for start of treatment was calculated form time of first presentation to hospital (day 0) till the first day of start of definitive first treatment for breast cancer. The investigator labelled delay in treatment if it was initiated later than 62days .

The questionnaire inquired about the symptoms, date of presentation of the first symptoms, date of first reporting to hospital, reasons for the delayed presentation.

All patients who were admitted and underwent pre anesthesia assessment underwent COVID testing according to the protocol. If the patient turned out COVID positive, their symptoms were noted and the COVID team (infectious disease department) was notified. The quarantine protocol at investigating hospital was, complete isolation for 14 days with one PCR-negative report after completing quarantine, with no residual respiratory symptoms of cough, fever, and shortness of breath. This protocol was followed for all elective breast surgery patients admitted in the hospital. All COVID-positive patients underwent the same treatment protocol as non-COVID patients with regards to management of breast cancer. Patients with early breast cancer (upto stage 2A) underwent modified radical mastectomy/breast conservative surgery first, followed by chemotherapy/radiotherapy, locally advanced cases (stage 2B and above) had neo-adjuvant treatment first followed by surgery, and advanced cases(stage 4/metastatic) underwent palliative treatment.

All the data obtained were analyzed using IBM SPSS 23.0. Descriptive statistics like age were presented as range and means. Categorical data were analyzed using fisher exact test and t-test was applied to numerical data. In all cases, a 95% confidence interval was used and p value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer confirmed on histo-pathological examination

Exclusion Criteria:

* Patients who had already had their surgery pre covid (December 2019)

Ages: 25 Years to 71 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer incidence is more in females as compare to male population
Study Population: Patient's data of all operated cases for suspicious lump breast (abnormal findings on ultrasound and mammogram, BIRAD III or above and abnormal FNAC results;C3 or above) from January1,2020 to 31 January 2021was retrieved. Out of these only those patients were included in whom the diagnosis of breast cancer was confirmed on histo-pathological examination. Patients who had already had their surgery pre covid (December 2019), were excluded. Data were collected on standard pre-designed questionnaire and from paper documents retrieved from patient records.
  All patients who were admitted and underwent pre anesthesia assessment underwent COVID testing according to the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Duration of delay in presentation to hospital | 18 months
  It was time counted from the day when the participant first felt breast symptom on self assessment or during diagnostic workup and than presented for the first time to hospital for diagnostic or treatment workup purpose
Duration of delay in definitive treatment | 18 months
  It was counted from the day of first presentation to hospital till the day of initiation of definitive treatment (chemo/surgery)
Cancer upstaging | 18 months
  It was assessed by reassessing the patient by comparison of disease stage on first time diagnostic workup results and than reassessing the stage of cancer during consecutive visits to hospital , and the effect of delay in treatment and presentation on cancer upstaging of participants related to covid 19 pandemic is evaluated .

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Ahmad Khan, MBBS, FCPS, Study Chair — PNS Shifa Hospital Karachi , HOD department of Surgery
Locations (1):
- Bahria University Medical and Dental College Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
impact of present covid 19 pandemic on presentation of breast cancer stage and disease upstaging status if patients are covid positive
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Gulzar F, Akhtar MS, Sadiq R, Bashir S, Jamil S, Baig SM. Identifying the reasons for delayed presentation of Pakistani breast cancer patients at a tertiary care hospital. Cancer Manag Res. 2019 Jan 29;11:1087-1096. doi: 10.2147/CMAR.S180388. eCollection 2019. PMID 30774437
- [Background] Khan MA, Shafique S, Khan MT, Shahzad MF, Iqbal S. Presentation delay in breast cancer patients, identifying the barriers in North Pakistan. Asian Pac J Cancer Prev. 2015;16(1):377-80. doi: 10.7314/apjcp.2015.16.1.377. PMID 25640384
- [Background] Vuagnat P, Frelaut M, Ramtohul T, Basse C, Diakite S, Noret A, Bellesoeur A, Servois V, Hequet D, Laas E, Kirova Y, Cabel L, Pierga JY; Institut Curie Breast Cancer and COVID Group; Bozec L, Paoletti X, Cottu P, Bidard FC. COVID-19 in breast cancer patients: a cohort at the Institut Curie hospitals in the Paris area. Breast Cancer Res. 2020 May 28;22(1):55. doi: 10.1186/s13058-020-01293-8. PMID 32460829
- [Result] Elghazawy H, Bakkach J, Zaghloul MS, Abusanad A, Hussein MM, Alorabi M, Eldin NB, Helal T, Zaghloul TM, Venkatesulu BP, Elghazaly H, Al-Sukhun S. Implementation of breast cancer continuum of care in low- and middle-income countries during the COVID-19 pandemic. Future Oncol. 2020 Nov;16(31):2551-2567. doi: 10.2217/fon-2020-0574. Epub 2020 Jul 27. PMID 32715776